CLINICAL TRIAL: NCT05233384
Title: Genomics of Fibrin Clot Structure in Patients With Constitutional Dysfibrinogenemia
Acronym: GENDYSFIB
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 LEBRETON; 2021-A00745-36 (Other: 2021-A00745-36)
Record Dates: First submitted 2022-01-06; First posted 2022-02-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Hereditary Dysfibrinogenemia
Keywords: Hereditary Dysfibrinogenemia; Fibrin clot; Polymorphism
MeSH Terms: conditions — Dysfibrinogenemia, Congenital | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hereditary dysfibrinogenemia: Patient, male or female, aged over 18, with confirmed hereditary dysfibrinogenemia
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — For each patient included, this study will involve the collection of 20 ml of blood during a blood test carried out as part of routine care. One EDTA tube (4,5 ml) will be withdrawn and frozen for genetic testing. 15 ml of citrated blood sample (3 to 5 tubes, depending on the used tubes) are necessary for the study of fibrin clot structure. Citrated tubes will be double centrifugated and frozen (-80°C) according to "Groupe Français d'Études sur l'Hémostase et la thrombose" guidelines (centrifugation protocol: 1500 to 2000g at least 15min, or 2000 to 2500g at least 10min with an intermediate decantation).

SUMMARY:
Hereditary dysfibrinogenemia results from monoallelic mutation in one of the fibrinogen genes (FGA, FGB, FGG). The spectrum of molecular abnormalities is broad, leading to several subtypes of coagulation disorders with specific biological and clinical features. The correlation between the genotype and the phenotype is poor, and the clinical course of patients, from major bleeding to recurrent thromboses, is unpredictable. Fibrin clot structure is a determinant of the risk of thrombosis in cardiovascular diseases. In all individuals, fibrin networks define the propensity of clot to be more resistant to removal or, on the contrary, susceptible to fragmentation leading to bleeding complications. Besides fibrinogen variants, other relatively common genetic polymorphisms in coagulation and fibrinolytic pathways may affect the fibrin clot structure and therefore act as modifiers of the blood clot function.

In this proposal, the investigators will analyze properties (polymerization, fibrinolysis, viscoelastic properties, permeation) and ultrastructure (size, number, packaging, architecture of fibrin fiber by confocal microscopy and scanning electron microscopy) of plasma-based clots in relation to the presence of genetic modifiers (polymorphisms). Polymorphisms will be detected using a whole exome sequencing (WES) in a selected panel of genes of the coagulation and fibrinolytic pathways. The gene panel of 28 genes will include the three fibrinogen genes plus 25 potential modifier genes including F5, F2, PAI-1, PROCR and MTHFR. The overall clot phenotype will be correlated to the presence of prothrombotic polymorphisms and to the patient's clinical phenotype. The investigators plan to include about 100 patients with dysfibrinogenemia. The combination of integrative hemostasis models with genetic dataset will provide a global view of the patient's individual hemostatic profile. This may allow to better predict the clinical outcome and help provide a more personalized therapeutic strategy and precision medicine. In addition, the development of models allowing a reliable global assessment of fibrin clot architecture will be the basis for further research in other acquired diseases involving thrombotic or bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed hereditary dysfibrinogenemia
* Able to give his/her informed consent to participate
* Affiliated to the French Health insurance

Exclusion Criteria:

* Refusal to participate
* pregnant and breastfeeding women,
* protected adults (individuals under guardianship by court order),
* adults deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with confirmed hereditary dysfibrinogenemia
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
relation between the genetic polymorphisms and the main parameters of each different tools evaluating the ultrastructure of fibrin clot | at the end of the inclusion period
  High quality genomic DNA will be purified using standard procedures and quantified using the Thermo Fisher Qubit fluorometric quantification. Whole exome sequencing will be performed at the Health 2030 Genome Center, Campus Biotech, Geneva using IDT Research Exome Reagents, multiplexing 12 samples during library preparation, for a mean coverage of 70x

SECONDARY OUTCOMES:
relation between the genetic polymorphisms and the clinical phenotype of patients with dysfibrinogenemia (thrombotic and/or bleeding phenotype) | at the end of the inclusion period
relation between the main parameters of ultrastructure of fibrin clot properties and the clinical phenotype of patients with dysfibrinogenemia | at the end of the inclusion period

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien LEBRETON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (7):
- France (7):
  - CHU clermont-ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU de Lille, Lille
  - CHU Montpellier, Montpellier
  - CHu Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Tours, Tours